CLINICAL TRIAL: NCT05047393
Title: Effect of Vitamin D Level on Pain Type in Coccygodynia
Brief Title: Vitamin D Level and Pain Type in Coccygodynia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cumhuriyet University (Other)
Responsible Party: Principal Investigator, Emel Güler, Associate Professor, Cumhuriyet University
Other Study IDs: 2021-06/21
Record Dates: First submitted 2021-08-31; First posted 2021-09-17 (Actual); Last update posted 2021-09-27 (Actual); Status verified 2021-09

CONDITIONS: Coccyx Disorder; Neuropathic Pain; Nociceptive Pain; Vitamin D Deficiency
Keywords: Coccyx; Nociceptive Pain; Neuropathic Pain; Chronic pain; Vitamin D Deficiency
MeSH Terms: conditions — Neuralgia; Nociceptive Pain; Vitamin D Deficiency; Chronic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples Without DNA — Venous blood samples will be obtained from the patients. Vitamin D level will be determined from blood samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Coccygodynia group: 51 patients with a diagnosis of coccygodynia will be included in the study.
  Interventions: Other: Current blood vitamin D level and painDetect questionairre score will be detected

INTERVENTIONS:
Other: Current blood vitamin D level and painDetect questionairre score will be detected — PainDETECT neuropathic pain questionnaire will be used to evaluate the presence of nociceptive, mixed and neuropathic pain in patients. Patients with a total questionnaire score of 12 or less are considered nociceptive pain without a neuropathic pain component. If the total score is in the range of 13-18, the result is uncertain, but it is accepted that the neuropathic component can be found in the mixed type, and in the scores of 19 and above, it is accepted that the neuropathic pain component is present. Patients with previously obtained and finalized vitamin D levels < 20 ng/mL, 20-30 ng/mL, and ˃30 ng/mL will be grouped as deficiency, insufficiency and normal, respectively.

SUMMARY:
Coccygodynia is a painful clinical picture of the sacrococcygeal region.Pain in coccygodynia may be somatic, neuropathic or mixed. There are many studies that emphasize the relationship between vitamin D deficiency and pain.In this study, it is aimed to investigate the severity and type of pain, as well as the effect of vitamin D level on pain in patients with coccygodynia

DETAILED DESCRIPTION:
There are different types of pain in coccygodynia. Patients may suffer from e somatic, neuropathic or mixed pain.Vitamin D plays an important role in the pathophysiology of pain. Vitamin D inhibits NO synthase (iNOS) in microglia and astrocytes. The importance of this is that nitric oxide (NO) is an important molecule in the development of neuropathic pain. NO production contributes to the maintenance of pain hypersensitivity. NO causes central sensitization and mechanical allodynia by increasing spinal cord posterior horn N-methyl-D-aspartate (NMDA) receptors.In the literature, it has been reported that low vitamin D level is associated with the severity of neuropathic pain in postherpetic neuralgia, diabetic neuropathy, rheumatoid arthritis and carpal tunnel syndrome, which cause neuropathic pain development.

Based on the above-mentioned data, in this study, I aimed to investigate the severity and type of pain, as well as the effect of vitamin D level on pain in patients with coccygodynia. Within the scope of the study, 51 patients with a diagnosis of coccygodynia will be recruited. Patients' age, gender, body mass index, duration of symptoms, etiology of coccycodynia, pain severity, pain type and blood vitamin D level will be recorded. Pain assessment (for discrimination between nociceptive, mixed and neuropathic pain) will be done with the painDETECT questionairre. Pain severity will be evaluated with Visual Analog Scale (VAS). Those with vitamin D levels < 20 ng/mL, 20-30 ng/mL, and ˃30 ng/mL will be grouped as deficiency, insufficiency and normal, respectively.The data will be entered into the SPSS (version: 22.0) IBM SPSS statistical package program. Arithmetic mean, standard deviation, min-max, median values will be given in the data obtained by measurement. Percentage and frequency distribution will be given in the data obtained by counting. In statistical evaluations, parametric tests will be used for normally distributed data, and non-parametric tests will be used for data not normally distributed. Relationships will be compared according to the Pearson or Spearman correlation coefficient. Chi-square test will be applied to categorical data. P<0.05 will be considered significant.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with coccygodynia
* 18-70 years old
* Having a vitamin D level determined
* Agreement to take part in the study.

Exclusion Criteria:

* Presence of known polyneuropathy,
* Presence of diabetes mellitus, renal failure, thyroid diseases
* Taking vitamin D replacement therapy,
* Using any of the medications used in the treatment of neuropathic pain such as duloxetine, pregabalin, gabapentin and tramadol, Having undergone an interventional procedure for coccygodynia within 3 months before the evaluation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who applied to Sivas Cumhuriyet University Faculty of Medicine Physical Therapy and Rehabilitation clinic between 01/08/2021 and 28/02/2022 and were diagnosed with coccygodynia and had their vitamin D levels checked will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 51 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-02-28 (Estimated); Study Completion 2022-02-28 (Estimated)

PRIMARY OUTCOMES:
Neuropathic pain in coccygodynia | The study will be completed in 7 months.
  PainDETECT neuropathic pain questionnaire will be used to evaluate the presence of neuropathic pain in patients.The questionnaire score ranges from 0-35 points, and a score of 19 and above indicates the presence of neuropathic pain.
Vitamin D level in coccygodynia | The study will be completed in 7 months.
  Vitamin D level of the patients registered in the hospital system will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Emel Güler, MD, Principal Investigator — Cumhuriyet University
Locations (1):
- Emel Guler, Sivas, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yesil H, Sungur U, Akdeniz S, Gurer G, Yalcin B, Dundar U. Association between serum vitamin D levels and neuropathic pain in rheumatoid arthritis patients: A cross-sectional study. Int J Rheum Dis. 2018 Feb;21(2):431-439. doi: 10.1111/1756-185X.13160. Epub 2017 Aug 31. PMID 28857474
- See also: Association between serum vitamin D levels and neuropathic pain in rheumatoid arthritis — https://pubmed.ncbi.nlm.nih.gov/28857474/